CLINICAL TRIAL: NCT05537090
Title: A Single Center, Open-label, 3-period Fixed-sequence, Phase I Clinical Study to Evaluate the Effect of BV100 on the Pharmacokinetics of Midazolam and Its Metabolite 1-hydroxymidazolam in Healthy Volunteers
Brief Title: A Study to Assess Effect of BV100 on the Pharmacokinetics of Midazolam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVersys AG (Industry)
Collaborators: Clinical Research Units Hungary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BV100-005
Record Dates: First submitted 2022-09-07; First posted 2022-09-13 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: This is an open-label, 3 period fixed-sequence, Phase 1 clinical study to evalu-ate the effect of multiple doses of BV100 on the Pharmacokinetics on midazo-lam and its metabolite 1-hydroxymidazolam in healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BV100 Plus Midazolam (Experimental): A total 2 doses of midazolam and 9 doses of BV100 will be administered to each participant per specified dosing schedule
  Interventions: Drug: BV100; Drug: Midazolam

INTERVENTIONS:
Drug: BV100 — Rifabutin for Infusion
Drug: Midazolam — Syrup for oral administration

SUMMARY:
To evaluate the effect of repeated doses of intravenous BV100 on the pharma-cokinetics of midazolam and 1-hydroxymidazolam.

DETAILED DESCRIPTION:
A single center, open-label, 3-period fixed-sequence, Phase I clinical Study to Evaluate the Effect of BV100 on the Pharmacokinetics of Midazolam and its metabolite 1-hydroxymidazolam in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who were able to understand and follow instructions during the study.
2. Subjects who signed informed consent.
3. Male subjects ≥18 and ≤55 years of age; female subjects ≥18 and ≤55 years of age of nonchildbearing potential defined as follows:

   * Female subjects 50 years of age or older, in menopause for 24 con-secutive months and not receiving any hormone replacement therapy within 24 months prior to inclusion into the study
   * Female subjects who underwent surgical sterilization
   * Female subjects who underwent hysterectomy
   * Female subjects with documented premature ovarian failure
4. Weight within a BMI range of 19.0-30.0 kg/m2.
5. Estimated glomerular filtration rate (eGFR) according to the CKD-EPI: ≥90 mL/min (normal renal function)
6. Healthy subjects had to be in a good health in the opinion of the study phy-sician, as determined by medical history, ECG, vital signs, physical examina-tion, and clinical laboratory tests.
7. Having had no febrile or infectious illness for at least 14 days prior to dos-ing.
8. The subject was available to complete the study.
9. The subject was complying with the restrictions and requirements of the protocol and, in the opinion of the study physician, was able to complete the study.

Exclusion Criteria:

1. Unwilling or unable to give informed consent.
2. As a result of the medical screening process, the study physician considered the subject unfit for the study.
3. Pregnant or lactating women or men with female partners who are lactating or are pregnant.
4. Known or suspected history of hypersensitivity to rifabutin or excipients or to drugs of a similar chemical class including rifampicin, rifapentine, rifaximin; history of allergic reactions leading to hospitalisation or any other allergic con-ditions (including drug allergies, asthma, eczema, anaphylactic reactions but excluding untreated, asymptomatic, seasonal allergies) which the Investigator considers may affect the safety of the subject and/or outcome of the study.
5. History of antibiotic associated diarrhoea within the last year.
6. Volunteers with ECG abnormalities (history, or evidence of second-degree heart block of Mobitz type II, third degree heart block, or any abnormality con-sidered relevant by the Investigator), QTcF > 450 ms, PR > 200 ms, or QRS duration > 110 ms.
7. Supine systolic blood pressure > 140 mmHg or < 90 mmHg or diastolic blood pressure > 90 mmHg or < 50 mmHg at Screening or Day 1 prior to dos-ing (any abnormal blood pressure results may be repeated once and if the re-peat result is within the normal range, it is not considered to have met the ex-clusion criterion). Pulse rate > 90 or < 50 beats per minute at Screening or Day 1 prior to dosing.
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and creatinine, above the ULN at Screening. Any abnor-mal value of these parameters may be repeated during screening period and if the repeat result is within the laboratory reference range, it is not considered to have met the exclusion criterion.
9. Screening values other than AST, ALT, ALP, creatinine, for haematology, biochemistry, or urinalysis must not exceed the reference range. Minor devia-tions from normal are allowed, if they are not clinically significant.
10. Leucocytes or neutrophils or lymphocytes below the lower limit of the ref-erence range.

11 History of symptomatic, chronic or recurrent infection (e.g. nausea, vomit-ing, diarrhoea, infection with fever) or any viral (including symptomatic herpes zoster), bacterial (including upper respiratory infection), fungal (non-cutaneous) or parasitic infection within 30 days prior to admission to the clini-cal unit.

12. A positive pre-study serology test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV)-1 and/or 2 antibodies.

13. Positive Coronavirus (SARS-CoV-2) rapid test and PCR (upon Check-in on Day -1) 14. A positive pre-study drug/alcohol screen. 15. History of epilepsy, other neurological disorders, or neuropsychiatric con-ditions.

16. History of seizures. 17. Volunteers who have received any prescribed systemic or topical medica-tion within 4 weeks of the first dose administration.

18. Subjects who had used any non-prescribed systemic or topical medication (including herbal remedies) or megadose vitamins (i.e. 20 to 600 times the rec-ommended daily supplement dose) within 7 days prior to dosing, unless in the opinion of the study physician the medication did not interfere with the study procedures or compromise safety.

19. Volunteers who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration.

20. Regular use of any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to the first admission to the clinical unit.

21. Volunteers who have participated in a clinical study involving administra-tion of an investigational drug (new chemical entity) within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (which-ever is longer).

22. Volunteers who consume more than 21 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 30 mL of 40% of alcohol by volume distilled spirits).

23. Excessive consumption of caffeine- or xanthine-containing food or bever-ages (> 5 cups of coffee a day or equivalent) or inability to stop consuming from 48 hours prior to study treatment administration.

24. Subjects who smoked more than 10 cigarettes a day. 25. Any use of drugs-of-abuse or alcohol abuse within 2 years prior to the first admission to the clinical unit.

26. Inability to understand or communicate reliably with the Investigator or considered by the Investigator to be unable to or unlikely to co-operate with the requirements of the study.

27. Any other conditions or factors which in the opinion of the Investigator may interfere with study conduct. Failure to satisfy the Investigator of fitness to participate for any other reason.

28. Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days prior to the first admission to the clinical unit.

29. Inability to refrain from using soft contact lenses starting from administra-tion of study treatment until follow-up visit.

30. Volunteers who are study site employees or immediate family members of the study site or Sponsor employee.

31. Contraindications related to midazolam: Hypersensitivity to the active sub-stance(s) or to any of the excipients, Severe hepatic impairment, Severe res-piratory failure or acute respiratory depression, Myasthenia gravis, Sleep ap-nea, Anatomical respiratory impairment or lung diseases. Note: as per Midazo-lam smpc "Pharmacokinetic interactions with CYP3A4 inhibitors or inducers are more pronounced for oral as compared to oromucosal or parenteral midazo-lam as CYP3A4 enzymes are also present in the upper gastrointestinal tract. Hence, a careful monitoring of the clinical effects and vital signs is recom-mended during the use of midazolam with a CYP3A4 inhibitor even after a single dose".

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of repeated doses of intravenous BV100 on the pharmacokinetics of midazolam | 0 (predose) up to 24 hours postdose on Day 1 and Day 7
  Maximum Observed Plasma Concentration (Cmax) of Midazolam
To evaluate the effect of repeated doses of intravenous BV100 on the pharmacokinetics of midazolam | 0 (predose) up to 24 hours postdose on Day 1 and Day 7
  Area Under the Plasma Concentration-Time Curve (AUC) of Midazolam
To evaluate the effect of repeated doses of intravenous BV100 on the pharmacokinetics of 1-hydroxymidazolam | 0 (predose) up to 24 hours postdose on Day 1 and Day 7
  Maximum Observed Plasma Concentration (Cmax) of 1-hydroxymidazolam
To evaluate the effect of repeated doses of intravenous BV100 on the pharmacokinetics of 1-hydroxymidazolam | 0 (predose) up to 24 hours postdose on Day 1 and Day 7
  Area Under the Plasma Concentration-Time Curve (AUC) of 1-hydroxymidazolam

SECONDARY OUTCOMES:
To evaluate the safety, and tolerability in healthy volunteers receiving multiple intravenous doses of BV100 with and without midazolam | 26 days
  Number of Participants with Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Geza Lakner, Principal Investigator — Clinical Research Units Hungary
Locations (1):
- CRU Hungary Kft., Early Phase Unit, Kistarcsa, Hungary

IPD SHARING:
Plan to Share IPD: No